CLINICAL TRIAL: NCT06160063
Title: The Effect of Educational Play on Diabetes Acute Complications and Health Literacy in Children: A Randomized Controlled Study
Brief Title: Diabetes Acute Complications and Health Literacy in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Fatma Yeşil, llecturer, University of Yalova
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023
Record Dates: First submitted 2023-01-15; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Childhood; Diabetes; Health Literacy
Keywords: Childhood; Diabetes; Health Literacy; Social Learning Theory; Board Game
MeSH Terms: conditions — Diabetes Mellitus | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: randomized control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): It is planned to meet with the experimental group 3 times in total. In the first interview, first of all, "Diabetes Child Diagnosis Form" and "Diabetes Health Literacy Scale for Acute Complications in Children" will be applied. Then the diabetes health literacy board game will be played. For this, groups of 4 will be formed and care will be taken to ensure that children of similar age groups are together while forming groups. In the clinic, they will be asked to play a diabetes health literacy (DISOY) board game in a quiet, bright room, a room with a table and 4 chairs. DISOY board game averages 45-60 minutes. and the first meeting will end here. Each child will be given one game to play with their parents at least twice at home.
  The second interview will be provided 1 month after the first interview. The third interview will be held in the third month. Data collection forms will be filled out again at each interview.
  Interventions: Behavioral: Education intervention
- control (No Intervention): control group; It is planned to meet with the control group 3 times in total. In the first, second and third interviews, only the data collection forms will be filled by the children.
  After collecting all the data of the experimental group, a board game will be given to the parents and children in the control group.

INTERVENTIONS:
Behavioral: Education intervention — Board game was created in line with current literature. In each interview, it is expected that the child's negative behaviors will be transformed into positive behaviors.
  Arms: Experimental group

SUMMARY:
In this study, in which education on acute complications of type 1 diabetes is planned with board games based on Bandura's social learning theory, children can indirectly learn common points that they may hear about acute complications of diabetes by watching board games of other group members. In line with this theory, children's knowledge needs regarding acute complications of diabetes can be determined, and interventions can be planned to meet the determined needs of children. Thus, the level of knowledge of diabetes health literacy for acute complications of diabetes can be increased.

This study will be carried out in a randomized controlled manner to evaluate the effect of educational play in children on acute complications of diabetes and health literacy.

DETAILED DESCRIPTION:
This study was conducted to determine the Turkish validity and reliability of the "Health Literacy Scale for Acute Complications of Type 1 Diabetes for Children (8-12 Years)" and to provide a diabetes health literacy box game to 8-12 school age children diagnosed with Type 1 diabetes. It will be carried out in two stages in order to evaluate the effect of educational games on acute complications of diabetes and health literacy in children.

In the first stage of the research, a general screening methodological method will be carried out to determine the current situation by quantitative analysis of the data obtained with the "Health Literacy Scale for Acute Complications of Type 1 Diabetes for Children (8-12 years)".

In the second stage; Randomly determined intervention and control groups will be applied to the intervention and control groups in a quasi-experimental type at the pre-test and the 1st and 3rd months after the training.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes age is at least one year
2. Regular attendance to the three-month routine outpatient clinics
3. Not having any other disease accompanying diabetes
4. The child is between 8-12 years old

Exclusion Criteria:

1. Children not coming to the given appointment
2. Children who do not play the diabetes health literacy (DISOY) board game at home

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Validity and reliability of the "Health Literacy Scale for Acute Complications of Type 1 Diabetes for Children (8-12 Years)" in Turkish | 6 month
  The Turkish validity and reliability of the "Health Literacy Scale for Acute Complications of Type 1 Diabetes for Children (8-12 Years)" was carried out.
  Scale items will be created by the researcher.
  The scale items will be presented to expert opinion and experts will be asked to evaluate the scale according to the Davis (1992) technique. Items that need to be revised will be reviewed and the final version of the scale will be created. Children who score higher on the scale will indicate a higher level of diabetes health literacy. The scale developed within the scope of the research will be filled in by children with diabetes themselves.
Evaluation of Literacy Scale for Acute Complications of Diabetesfor Children with Type 1 Diabetes (8-12 years) | Baseline, 4 weeks ve 12 weeks after randomization
  The diabetes health literacy of children with type 1 diabetes aged 8-12 years who participated in our research was evaluated with the "Literacy Scale for Acute Complications of Diabetes for Children with Type 1 Diabetes (8-12 years)" scale. The scale was applied to the participants at the first meeting. Then, diabetes education was given to the participants through games. The scale was re-administered to the participants 1 and 3 months after the training. Participants were advised to play the game at least twice between follow-ups.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul İl Sağlık Müdürlüğü, Istanbul, Turkey (Türkiye)